CLINICAL TRIAL: NCT03590301
Title: Third Ward Wellness Study for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Tracey Ledoux, Associate Professor, University of Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001076
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know whether they are in the control or experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FUNPALs Playgroup (Experimental): Based on Self-Determination Theory, the FUNPALs Playgroup will enable and inspire parents to encourage their children to improve their diet and activity behaviors through general authoritative parenting, structured feeding practices, and a healthy home environment. Parents and toddlers will participate in the FUNPALs Playgroup together where they will be led through a series of open but structured activities including free play, exercise, snack preparation, discussion, singing, and yoga stretches.
  Interventions: Behavioral: FUNPALs Playgroup
- Healthy Toddlers Parent Group (Active Comparator): The goal of the Healthy Toddlers Parent Group is to deliver the same nutrition and activity messages to parents as those delivered in the FUNPALs Playgroup. In the Healthy Toddlers Parent Group, parents (without children) will meet in groups to receive information on nutrition and activity as it relates to their toddlers and they will engage in a discussion around how they do or can implement these behaviors. No experiential learning, children, play, or parenting instruction will be included in this control condition.
  Interventions: Behavioral: Healthy Toddler Parent Group

INTERVENTIONS:
Behavioral: FUNPALs Playgroup — Based on Self-Determination Theory, the FUNPALs Playgroup aims to enable and inspire parents to improve their toddlers dietary intake and physical activity habits through authoritative parenting, structured feeding practices, and a healthy home environment. Playgroups will include open but structured experiential learning activities, free play, and instruction/discussion.
  Other Names: experimental group
  Arms: FUNPALs Playgroup
Behavioral: Healthy Toddler Parent Group — The parent class will serve as our instruction only control group. Parents in this class will receive information about nutrition and activity recommendations regarding their toddler age children and will discuss it in a group with other parents. No experiential learning activities, information about parenting, or children will be involved in this class.
  Other Names: control group
  Arms: Healthy Toddlers Parent Group

SUMMARY:
The Third Ward Wellness Study aims to pilot test a wellness program for families with toddler age children. Participants will be recruited from the Third Ward neighborhood in Houston, TX and then randomly assigned to one of two wellness programs. The goal of both programs is to enable and inspire parents to help their toddler age children develop healthy habits that will stay with them through life. Participating families will complete an assessment batter before and after the program. Both programs will meet once per week for 10 weeks.

DETAILED DESCRIPTION:
Dietary and activity habits begin to develop in early childhood. Parents have the most influence on children's health behaviors at this age. Many parents, particularly those from lower income and underserved areas may benefit from programs to inspire and enable them to raise their toddler age children with good health habits. The experimental group was developed to help parents instill healthy habits in their children through a healthy home environment. This study will pilot test the experimental group among parent-toddler dyads residing in Greater Third Ward neighborhoods, where > 80% of the residents are AA or Hispanic and 35%-54% have annual household incomes <$25,000. The aims are to ascertain 1) recruitment and retention barriers and facilitators, 2) treatment success barriers and facilitators, and 3) the estimated effect sizes of outcomes to inform a fully powered RCT. The exploratory hypotheses are that compared to those in the control group, parents in the experimental group will have greater increases in positive parenting skills (Comprehensive General Parenting Questionnaire), and toddlers will have greater increases in indicators of a healthy home environments, diets and activity habits (MVPA, sedentary activity, and sleep).

ELIGIBILITY:
Inclusion Criteria:

Parents need to be...

* The legal custodian of a toddler,
* At least 18 years,
* Able to make food decisions in the home,
* Have access to a phone at home,
* Be fluent in English Toddlers need to be...
* Between 12 and 36 months of age
* Be able to walk.

Exclusion Criteria:

* Adults unable to consent for themselves and their child,
* Parents or toddlers who have mental or physical health conditions that would prevent them from fully engaging in activities of the program (e.g., reliance on feeding tube).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Comprehensive General Parenting Questionnaire | Baseline and immediate post intervention
  This 69-item measure of general parenting will assess changes in domains of positive parenting (i.e., authoritative parenting): nurturance, structure, and behavioral control.

SECONDARY OUTCOMES:
Structure Feeding Practices (Savage et al., 2017) | baseline and immediate post intervention
  This 22 item measure will assess limiting exposure to unhealthy foods and establishing mealtime routines
Home environment | baseline and immediate post intervention
  a phone interview will assess home availability of foods, physical activity resources, screen media devices, and sleep conditions as well as social norms and family policies regarding meals, active play, sleep, and screen media
Toddler fruit and vegetable intake | Baseline and immediate post intervention
  Dermal reflectance spectrometry (Veggie Meter (R), Longevity Link Corp) will used to assess skin carotenoid levels of the toddlers. Skin carotenoid levels reflect dietary intake of carotenoids, which are pigments found in many fruit and vegetables
Toddler dietary intake | baseline and immediate post intervention
  The Kids Bites Food Frequency Questionnaire (Aguilar et al., 2014) will assess consumption of snack foods, sugar, sweetened beverages and fruit and vegetables. Parents will complete this measure for their children.
Child sedentary, moderate to vigorous, and sleep activity | Baseline and immediate post intervention
  Toddlers will wear the GT3X+ Actigraph (Pensacola, FL) for 8 consecutive days at baseline and immediate post. THe actigraph is a triaxial accelerometer that has been validated on toddler age children to measure activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Ledoux, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No